CLINICAL TRIAL: NCT04984564
Title: Cardiovascular Fellow-in-training Feedback on Virtual and Simulator-based Learning Experience During Covid-19 Pandemic in A Low to Middle Income Country
Brief Title: Cardiovascular Fellow-in-training Feedback on Virtual and Simulator-based Learning Experience in A Low to Middle Income Country
Status: Completed | Type: Observational
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Pirbhat Shams, Resident Physician, Co-Investigator, Aga Khan University Hospital, Pakistan
Other Study IDs: 2020-5030-10817
Record Dates: First submitted 2021-07-28; First posted 2021-07-30 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Educational Problems
Keywords: cardiovascular education, virtual education, simulator, LMIC

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None. As this was an observational study. — Observational study.

SUMMARY:
Virtual and simulatorbased learning is not widely available in LMIC. It is imperative to analyze feedback of CV fellow-in-training regarding this mode of learning before large scale implementation.

DETAILED DESCRIPTION:
COVID-19 pandemic has introduced us to a greater need of virtual learning platforms and has resulted in less clinical exposure for fellows-in-training. Virtual and simulatorbased learning is not widely available in LMIC. It is imperative to analyze feedback of CV fellow-in-training regarding this mode of learning before large scale implementation.

This was an observational study conducted between July-August 2020. A multicentered survey was conducted. Survey questionnaire was disseminated to FIT via Google Forms. The questionnaire contained total of 24 questions about virtual and simulator-based learning during the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Cardiovascular fellow-in-training currently under training at the institute.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All fellow in training who were enrolled in a cardiovascular post graduate training program were invited to fill in GoogleForm survey.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Feedback of individual fellow in training on virtual and simulator based learning. | Survey was conducted from august to july 2020. Subjects had two month period to respond.
  Fellows responded to survey questions.

CONTACTS AND LOCATIONS:
Overall Officials: Pirbhat Shams, MBBS, Principal Investigator — The Aga Khan University Hospital
Locations (1):
- Pirbhat Shams, Karachi, Outside US and Canada, Pakistan

IPD SHARING:
Plan to Share IPD: No